CLINICAL TRIAL: NCT03661853
Title: Effect of CBT Microinterventions on Mechanisms of Behavior Change Among Adults With AUD: Using Eye Tracking to Measure Pre-Post Cognitive Control, Stimulus Salience, and Craving
Brief Title: Effect of CBT Microinterventions on Mechanisms of Behavior Change Among Adults With AUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Epstein, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB ID: H00011382; 1R21AA025488-01 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: 4 arms: 3 CBT microinterventions + control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): This microintervention is intended to control for the effect of nonspecific therapy factors such as therapeutic alliance, time spent with a therapist, talking about alcohol, and/or effects related to assessment reactivity, and consists of 60 minutes of psycho-education on alcohol and drugs. The therapist will talk about historical and scientific information on different types of alcohol and drugs and will not overlap with CBT treatment. The participants will not be encouraged to personalize this information, make any behavioral changes, or do homework. The control does not have any active interventions that would specifically target or affect our outcome variables.
  Interventions: Behavioral: Control
- Functional Analysis (Experimental): Functional Analysis (FA) is a core intervention in Cognitive Behavioral Therapy (CBT) for AUD, and helps to "break the chain" of events (external and internal) that lead from cue (trigger) to alcohol use to consequences of use. The FA microintervention teaches the patient to think and behave in new, more controlled ways in response to triggers, to identify maladaptive, impulsive behavior chains and to replace them with more deliberate ones.
  Interventions: Behavioral: Functional Analysis
- Cognitive Restructuring (Experimental): Cognitive Restructuring of Thoughts About Alcohol (CR) is a core technique in CBT to help patients identify "automatic" (habituated) thoughts that happen quickly and are often not noticed, and change automatic thoughts occurring in response to alcohol triggers.
  Interventions: Behavioral: Cognitive Restructuring
- Dealing with Cravings (Experimental): Dealing with Cravings (DC) is designed to directly target the reward and arousal systems, helping the patient accept the nature of cravings as time limited and deflated by continued abstinence so that craving is no longer associated with urgency. DC also teaches skills to reduce cravings by conjuring images such as a spider floating in a glass of wine, or of older versions of oneself sitting alone and dejected in a bar. Distraction techniques and breathing skills to reduce physiological arousal occurring in response to alcohol cues are also taught.
  Interventions: Behavioral: Dealing With Cravings

INTERVENTIONS:
Behavioral: Control — 60 minute psycho-education on alcohol and drugs.
  Arms: Control
Behavioral: Functional Analysis — Component of standard CBT that helps to "break the chain" of events (external and internal) that lead from cue (trigger) to alcohol use to consequences of use.
  Arms: Functional Analysis
Behavioral: Cognitive Restructuring — CR is used to to help identify and change automatic, habituated thoughts that occur in response to alcohol triggers.
  Arms: Cognitive Restructuring
Behavioral: Dealing With Cravings — DC is used reduce cravings for alcohol by conjuring negative images associated with alcohol, teaching distraction techniques, and teaching breathing techniques to reduce physiological arousal.
  Arms: Dealing with Cravings

SUMMARY:
This proposed R21, Effect of CBT Microinterventions on Mechanisms of Behavior Change among Adults with AUD: Using Eye Tracking to Measure Pre-Post Cognitive Control, uses a translational team science approach to isolate and examine the effect of three different Cognitive Behavioral Therapy (CBT) interventions (functional analysis (FA), cognitive restructuring for alcohol related thoughts (CR), and dealing with cravings (DC)) on specific hypothesized mechanisms (cognitive control, stimulus salience, or craving/arousal, respectively).

DETAILED DESCRIPTION:
This R21 uses an innovative paradigm pairing a "microintervention" design with eye tracking laboratory tasks used successfully to show deficits of cognitive control over cocaine and nicotine cues, and to objectively measure stimulus salience and craving/arousal in response to alcohol cues. To achieve the study's two specific aims, participants with AUD will be assessed with antisaccade (to measure cognitive control) and attentional bias (to measure stimulus salience and pupil diameter) eye tracking tasks.

Specific Aim 1. To isolate and preliminarily assess the impact of specific CBT microinterventions on potentially malleable hypothesized mechanisms of change in drinking using a novel laboratory paradigm and conducted by a translational science team.

Specific Aim 2. To test specificity of CBT interventions' effect on particular Mechanisms of Behavioral Change, the investigators will test each microintervention's effects on all three purported mechanisms (as stated in "Brief Summary".)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Current Alcohol Use Disorder (AUD) Diagnosis
* Drank Alcohol within 60 days prior to telephone screen
* Able to read and understand English at the 7th grade education level

Exclusion Criteria:

* Participant diagnosed with Schizophrenia or Schizoaffective Disorder
* Participant has a head injury with symptoms in the last 30 days
* Current inpatient or outpatient treatment for AUD or Drug use Disorder (DUD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Changes in Drinking Behavior | Weekly for up to 3 weeks
  Changes in drinking behavior are measured by tracking eye movement patterns using antisaccade + attentional bias eyetracking tasks. Specifically, outcome mediators include changes in cognitive control (# of errors in antisaccade eye-tracking task), changes in stimulus salience (stimulus dwell time measurements), and changes in craving/arousal (pupil diameter changes in response to stimuli presentation.)

SECONDARY OUTCOMES:
Alcohol Use Questionnaire (AUQ) | Weekly for up to 3 weeks
  AUQ is an 8-item questionnaire that measures self-reported craving for alcohol. Item scores range from 1-7 and a total score, ranging from 8-56, is calculated by summing all values. Higher scores indicate greater craving.

OTHER OUTCOMES:
Barratt Impulsivity Questionnaire | Weekly for up to 3 weeks
  The Barratt is a 30-item questionnaire that measures self-reported general impulsivity. Item scores range from 1-4 and a total score, ranging from 30-120, is calculated by summing all values. There are three sub scales (Attentional, Motor, and Nonplanning) which are derived from individual items. Higher scores indicate greater attentional, motor, and nonplanning impulsivity and scores range from 8 to 32, 11 to 44, and 11 to 44, respectively.
Treatment Services Review | Given at Week 2 and Week 3 appointments out of 3 week program
  Interview assessing quantity and type of services received (e.g., health, psychological) outside of study intervention. Total scores are calculated by summing the number of outside services used. Total scores have a minimum of 0 and no maximum value.
Working Alliance Inventory Short Form | Week 2 appointment out of 3 week program
  12-item self-report measure of the therapeutic alliance. Total scales are calculated by summing all values. Values range from 1-7 with total scores ranging from 12 to 84. Higher scores indicate greater alliance.
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) | Measurement taken at baseline
  19 item self-report questionnaire assessing client readiness for change. An additional item assesses the client's motivation for coming to therapy. Item scores range from 1 to 5 and a total score, ranging from 19 to 95, is calculated by summing all values. There are three sub scales (Recognition, Ambivalence, and Taking Steps) which are derived from individual items. Higher scores indicate greater recognition, ambivalence and taking steps and scores range from 7 to 35, 4 to 20, and 8 to 40, respectively.
Use of Treatment Skills (UTS) | Week 3 appointment out of 3 week program
  UTS is an 18-item questionnaire that measures adherence to microintervention homework assigned at week 2 appointment. Item scores range from 0 to 4 and a total score, ranging from 0 to 72, is calculated by summing all values. Higher values indicate greater adherence to assigned homework.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Epstein, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Elizabeth E Epstein, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with investigators outside the core study team.